CLINICAL TRIAL: NCT02004834
Title: A Combination of Levobupivacaine and Lidocaine for Paravertebral Block in Breast Cancer Patients Undergoing Quadrantectomy Causes Greater Hemodynamic Oscillations Than Levobupivacaine Alone
Brief Title: Levobupivacaine and Lidocaine for Paravertebral Block Causes Greater Hemodynamic Oscillations Than Levobupivacaine
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Miroslav Župčić, Anesthesiology, Resuscitation and Intensive Care Medicine Specialist, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 260320131980
Record Dates: First submitted 2013-11-06; First posted 2013-12-09 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Tumors; Hypotension; Bradycardia
MeSH Terms: conditions — Breast Neoplasms; Hypotension; Bradycardia | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0,5% levobupivacaine with 2% lidocaine (Active Comparator): 7,0 ml.of mixture 0,5% levobupivacaine with 2% lidocaine are given per level Th2,Th3,Th4 for ultrasound guided paravertebral blocks in breast surgery
  Interventions: Drug: levobupivacaine
- 0,5% levobupivacine (Active Comparator): 7,0 ml. 0,5% levobupivacaine are given per level Th2,Th3,Th4, given for ultrasound guided paravertebral blocks in breast surgery
  Interventions: Drug: levobupivacaine

INTERVENTIONS:
Drug: levobupivacaine — Comparing: 0,5% levobupivacaine with 2% lidocaine
  Other Names: chirocaine

SUMMARY:
The purpose and the goal of this paper is to show whether the application of a combination of two local anesthetics, as opposed to the application of one local anesthetic at paravertebral block changes the hemodynamic variable. It is therefore a prospective randomized double- blind study, where we do a clinical trial in patients ASA(American Society of Anesthesiologists) 1 and 2 statuses between 18 and 80 years of age, using the ultrasound in plane technology.Upon arrival of patients in the unit for preparation procedures for anesthesia we set the ECG(electrocardiograph), noninvasive blood pressure, oxygen saturation, and arterial cannula in the radial artery After sterile washing of the dorsal surface, paravertebral space was identified with ultrasound using 8 Hz(hertz) linear transducer probe then needle position was confirmed with neurostimulation at the level of 2.0 - 5.0 mA(milliampere). When muscle contraction persisted at 0.4mA(milliampere), the anesthetic was applied in levels of Th 2, Th3, and Th 4 (7,0 milliliters per level). We applied the 0.5 % levobupivacaine and 2 % lidocaine, 7,0 milliliters of mixture per level in one group, while only 0.5 % levobupivacaine also 7,0 milliliters. by level in the second one. After that, the invasive hemodynamic monitoring was placed on patients and the induction with 1 % propofol 2-2.5 mg/kg.and Vecuronium 0,08 mg/kg. was performed with the application of supraglottic airway gel of appropriate size. The maintenance of anesthesia and sedation will be conducted with Propofol 1 % continuously ( 25-150 mcg / kg / min.)The measurements will be taken every 5 minutes during the first hour of the application of paravertebral block, then every 15 minutes during the second hour and if the operation takes more than two hours, the measurements are performed every 30 minutes. Postoperatively, invasive hemodynamic monitoring will be removed in post-anesthesia recovery room together with the arterial cannula and the patient will be sent to the hospital ward with non-invasive hemodynamic monitoring (blood pressure, pulse, saturation) until the termination of the blocks.Statistical methods, By comparing two target groups, we analysed the strength of the test with following assumptions: X2 difference test, the expected difference in variances in stroke volume between groups of 60%, α significance level of 0.05, and the minimum statistical test strength of 85%. The required total sample should include at least 80 patients, that is, 40 per group.Data will be presented in tables and graphs. Descriptive statistics of examined variables with appropriate measures of central tendency will be made. Smirnov -Kolmogorov test will assess the normality of data distribution. According to the received results, the appropriate parametric and / or nonparametric tests will be used. Comparisons of quantitative values between the two groups will be analyzed using the independent t-test or Mann-Whitney U test. Dependent values within each group will be analyzed using analysis of variance for repeated measures or Friedman test. Differences in categorical values will be analyzed by X2 test. The appropriate regression model will be made in order to predict the variability of stroke volume in which the dependent variable will be a variation of the stroke volume, while relevant clinical values will be taken as predictor variables. All P values smaller than 0.05 will be considered significant.

This research is to present the main results - the existence of the significant change in Stroke Volume Variation (SVV) between groups using invasive hemodynamic monitoring, the changes of Stroke Volume Variation(SVV) depending on the time from the application within groups, differences in volume compensation of crystalloids and colloids and the need for the application of vasoactive drugs. Furthermore, as a secondary results we will present the time to maximal block development, the duration of post operative analgesia, patient satisfaction and time needed for the full recovery from the block.

ELIGIBILITY:
Inclusion Criteria:

* ASA one and two status
* regular heart rhythm
* weight between 50 and 95 pounds

Exclusion Criteria:

* patient refusal
* coagulation disorder
* allergy to local anesthetics
* arrhythmias with or without valvular disease
* hypertension
* weight less than 50 pounds or more than 95 pounds

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Stroke Volume Variation(SVV)within and between groups of patients | 12 hours perioperative
  Determine which solution of local anesthetic with paravertebral block has a the most favorable effect with regard to the analgesic and hemodynamic effects.
  Stroke Volume Variation(SVV)will be expressed in percentage change.

SECONDARY OUTCOMES:
postoperative analgesic consumption | 12 hours
  Achieve satisfactory postoperative analgesia and thereby faster patient mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Ino Husedzinovic, PhD,MD, Study Chair — Clinical Hospital Dubrava, Head of Anesthesiology, Resuscitation and Intensive Care Medicine
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Background] Saito T, Den S, Cheema SP, Tanuma K, Carney E, Carlsson C, Richardson J. A single-injection, multi-segmental paravertebral block-extension of somatosensory and sympathetic block in volunteers. Acta Anaesthesiol Scand. 2001 Jan;45(1):30-3. doi: 10.1034/j.1399-6576.2001.450105.x. PMID 11152029
- [Background] Hara K, Sakura S, Nomura T. [Use of ultrasound for thoracic paravertebral block]. Masui. 2007 Aug;56(8):925-31. Japanese. PMID 17715684
- [Background] Garutti I, Olmedilla L, Cruz P, Pineiro P, De la Gala F, Cirujano A. Comparison of the hemodynamic effects of a single 5 mg/kg dose of lidocaine with or without epinephrine for thoracic paravertebral block. Reg Anesth Pain Med. 2008 Jan-Feb;33(1):57-63. doi: 10.1016/j.rapm.2007.07.009. PMID 18155058
- [Background] Kungys G, Rose DD, Fleming NW. Stroke volume variation during acute normovolemic hemodilution. Anesth Analg. 2009 Dec;109(6):1823-30. doi: 10.1213/ANE.0b013e3181ba41af. PMID 19923509
- [Background] Alhashemi JA, Cecconi M, della Rocca G, Cannesson M, Hofer CK. Minimally invasive monitoring of cardiac output in the cardiac surgery intensive care unit. Curr Heart Fail Rep. 2010 Sep;7(3):116-24. doi: 10.1007/s11897-010-0019-3. PMID 20623210
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Result] Batra RK, Krishnan K, Agarwal A. Paravertebral block. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):5-11. No abstract available. PMID 21804697
- [Result] Tahiri Y, Tran DQ, Bouteaud J, Xu L, Lalonde D, Luc M, Nikolis A. General anaesthesia versus thoracic paravertebral block for breast surgery: a meta-analysis. J Plast Reconstr Aesthet Surg. 2011 Oct;64(10):1261-9. doi: 10.1016/j.bjps.2011.03.025. Epub 2011 Apr 12. PMID 21486711